CLINICAL TRIAL: NCT07054359
Title: "HBV unIversal vs Point-Of-Care-based Antiviral treatMent to Prevent Mother-to-child Transmission"
Acronym: HIPOCAMP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ANRS 0562s HIPOCAMP
Record Dates: First submitted 2025-01-09; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: HBV Infection; Pregnancy
Keywords: Pregnancy; Mother to child transmission; Public health; Hepatitis B; Cluster-randomized controlled trial
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Intervention Model Description: A two-arm parallel cluster-randomized, open-label, non-inferiority trial will be conducted in five countries across two regions: sub-Saharan Africa (Cameroon, Ivory Coast, Togo) and Asia (Cambodia, Vietnam). The randomization (cluster) unit will be a primary health center (PHC) or a rural hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Universal strategy (Other): Pregnant women who test positive for HBsAg will initiate TDF preventive treatment on the same day of their visit. Their child/children will be enrolled in the study until 9 months.
  Interventions: Diagnostic Test: HBsAg RDT Women; Drug: Treatment by TDF; Other: Social sciences component; Diagnostic Test: HBsAg RDT Infants
- Selective strategy (Experimental): Pregnant women who test positive for HBsAg will be tested for HBcrAg RDT on the same day of their visit, and those who test positive will initiate TDF preventive treatment on the same date.Their child/children will be enrolled in the study until 9 months.
  Interventions: Diagnostic Test: HBsAg RDT Women; Drug: Treatment by TDF if HBcrAg RDT positive; Other: Social sciences component; Diagnostic Test: HBsAg RDT Infants

INTERVENTIONS:
Diagnostic Test: HBsAg RDT Women — HBsAg will be screened using finger-stick capillary blood during the ANC visit, simultaneously with the HIV test
Drug: Treatment by TDF if HBcrAg RDT positive — 300mg per day or 300 mg every 2 days (if créatinine clearance is 30-50ml/min)
  Arms: Selective strategy
Drug: Treatment by TDF — 300mg per day or 300 mg every 2 days (if créatinine clearance is 30-50ml/min)
  Arms: Universal strategy
Other: Social sciences component — The social sciences component only in Cambodia and Ivory Coast. 3 key sub-studies: i) a socio-economic and behavioral study ii) a health economic evaluation study, and iii) a health policy study.
  A mixed-methods approach will be used, including qualitative interviews and quantitative questionnaires among pregnant women and healthcare workers
Diagnostic Test: HBsAg RDT Infants — At 9 months, all infants will be tested for HBsAg; HBsAg-positive infants will undergo HBV DNA testing, and DBS will be collected for biobank storage.

SUMMARY:
To achieve global elimination of hepatitis B virus (HBV), it is crucial to eliminate HBV mother-to-child transmission (MTCT) by ensuring high coverage of birth dose vaccine and expanding the adoption of peripartum antiviral prophylaxis (PAP) by tenofovir. Current international guidelines require hepatitis B surface antigen (HBsAg)-positive pregnant women to undergo viral load (VL) quantification to identify those at high risk (VL ≥200,000 IU/mL) who should receive PAP. However, VL testing remains inaccessible in many low- and middle-income countries (LMICs), particularly in rural areas. Consequently, in the forthcoming guidelines, the WHO is going to issue a conditional recommendation for administering PAP to all HBsAg-positive women lacking access to VL testing. Although this universal strategy may appear promising for simplifying the diagnostic process, it may result in overtreating the majority of HBsAg-positive pregnant women, estimated at 85% in Africa and 70% in Asia, for whom birth dose vaccine is likely sufficient. Moreover, the real-world applicability of this strategy in LMICs has never been formally tested.

As an innovative alternative, the adoption of a rapid point-of-care test for hepatitis B core-related antigen (HBcrAg-RDT) is proposed to identify women eligible for PAP.This test requires only a drop of capillary blood, eliminating the need for electricity or centrifugation, and can provide a reliable result within 45 minutes. Compared to the universal strategy, HBcrAg-RDT strategy is expected to be less expensive and could prevent unnecessary tenofovir exposure for both women and their fetuses. Our aim is to establish the non-inferiority of the HBcrAg-RDT strategy, in comparison to the universal strategy, in terms of effectiveness, defined as the reduction in maternal VL at the time of childbirth, a main driver of the MTCT risk. This will be approached through a multidisciplinary framework integrating health economics, implementation science, and health policy analysis.

DETAILED DESCRIPTION:
I) Methodology and Study Design

The study combines two components:

I. Core Research Study Study Design Two-Arm Parallel, Cluster-Randomized Trial Design, Open-Label, Non-Inferiority Trial 1:1 Allocation Ratio 1:1 Arm 1: Intervention Group (Selective Strategy) HBsAg-positive women → Tested for HBcrAg RDT → TDF treatment if HBcrAg positive.

Arm 2: Control Group (Universal Strategy) HBsAg-positive women → Immediate TDF treatment

Clusters Randomization unit: Primary Health Centers (PHCs) or rural hospitals Total clusters: 80 (40 per group, 16 clusters per country)

Participants Total participants: 3200 HBsAg-positive women 1600 women per group → 640 women per country → 40 per cluster

Key eligibility criteria for clusters include:

* Rural or semi-rural location.
* No involvement in similar strategies
* No routine HBV DNA or HBeAg testing.
* Enough antenatal care visits to reach the target of 40 HBsAg-positive women in one year
* At least two nurses or midwives.
* HBV vaccination program in place
* Motivation to participate.

II. The Social Science component:

The social sciences component of the study will be conducted in only 2 countries (Cambodia and Ivory Coast) and includes three key sub-studies:

* The socio-economic and behavioral study aims to assess i) the acceptability of the two strategies by the healthcare workers involved in implementing the trial in the study sites and by the pregnant women who will participate in the trial and benefit from HBV PMTCT interventions, ii) the impacts of the strategies on health literacy, HBV knowledge, perceived health, treatment adherence and retention into care, iii) women experience related to HBV status disclosure and perceptions on HBV partner and children screening
* The health economic evaluation will analyze the strategies' costs, benefits, and cost-effectiveness, considering health and cost outcomes over the study period and the long term.
* The health policy study will evaluate the feasibility and sustainability of the strategies at the institutional level and explore political, institutional, and social factors that influence integrating the study results into national health policies.

A mixed-methods approach will be used, including qualitative interviews and quantitative questionnaires among pregnant women and healthcare workers.

Additionally, a qualitative assessment of the two strategies' acceptability, alongside a health policy analysis, will be conducted in Togo to enrich the study's contextual understanding. This initiative will also enhance the partner team's social science research capacity through targeted training and skill development in qualitative research for students and early-career researchers.

II) Intervention:

Medication: Tenofovir Disoproxil Fumarate (TDF); Administration Route: Oral Dosage: 300 mg/day or 300 mg every 2 days (if creatinine clearance is 30-50 ml/min)

Preventive treatment:

* Initiated during inclusion visit (if eligible for treatment in group 1, and for all in group 2)
* Continued until the 6-8 weeks postpartum visit Post-partum assessment and treatment At 3-month postpartum, all HBsAg-positive women will undergo a liver disease assessment at the closest district or provincial hospital. This assessment will include HBV DNA, HBeAg, HBcrAg-RDT, ALT/AST, platelet count, and liver ultrasound. Criteria for resuming treatment will follow the 2024 WHO guidelines. In case of TDF resumption, the treatment will be funded by the trial for 6 months, and the woman will be followed at a district or provincial hospital

III) Statistical methods

Core research study. The investigators predict that with the universal strategy, the proportion of women meeting the primary endpoint would be 78%. They chose a non-inferiority margin of 10% when comparing the HBcrAg-RDT strategy to the universal strategy. This indicates that a 68% success rate would be accepted for the same primary endpoint under the worst-case HBcrAg-RDT strategy.

They plan to recruit 40 HBsAg-positive women in each PHC. With a coefficient of variation between clusters of 0.143, derived from the assumptions, the trial requires 40 clusters per group, totaling 80 clusters of 40 HBsAg-positive women each, for 90% power at two-sided 5% (2.5% one-sided) significance to show non-inferiority within a margin of 10%.

Social Science quantitative data:

The sample size for the social science data is based on the proportion of women with good knowledge of hepatitis B, 90% power, two-sided 5% significance, and 20% loss to follow-up at the 9-month postpartum visit. Assuming 23% and 29% of women having good knowledge of hepatitis B at inclusion and the 9-month postpartum visit, respectively, overall for both strategies, with a correlation coefficient before-after of 0.15, 32 clusters (16 per country) of 40 women each (totaling 1280 participants) will be needed to show significant differences in the proportion of women with good knowledge of hepatitis B between inclusion and the 9-month postpartum visit (overall, considering both strategies together).

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old, or ≥ the legal age of majority as defined by each country, on the day of inclusion.
2. Pregnancy.
3. Intention to attend antenatal care visits in the Primary Health Center or the Rural Hospital
4. Living in an area covered by the Primary Health Center or the Rural Hospital on the start date of the trial
5. Positive HBsAg identified during the screening phase of the study
6. Free, informed, and written consent, signed by the person and the investigator at the latest on the day of inclusion and before any examination carried out as part of the study.

Exclusion Criteria:

1. HIV co-infection.
2. HBV treatment ongoing on the day of inclusion.
3. Having at least one of the following criteria indicatives of the third trimester of pregnancy:

   * Gestational Age-Based Exclusion:

   The reported gestational age is ≥28 weeks, based on the last menstrual period (LMP) if known.
   * Ultrasound-Based Exclusion:

   Fetal biometry (e.g., head circumference, femur length) on ultrasound suggests a gestational age of ≥28 weeks.
   * Fundal Height-Based Exclusion:

   Symphysis-fundal height (SFH) measurement of ≥ 28 cm which corresponds to approximately 28 weeks of gestation.
4. Severe gravid disease at inclusion, which poses a life-threatening risk to the mother and/or child
5. Any concomitant medical condition that, according to the clinical site investigator, would contraindicate participation in the study.
6. Concurrent participation in any other study (unless approved in writing by the Global Principal Investigators).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3200 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of HBsAg-positive women with HBV DNA <200,000 IU/mL at the time of delivery | Delivery
  The primary endpoint will be the percentage of HBsAg-positive women who present at healthcare facilities for delivery and have an HBV DNA <200,000 IU/mL at the time of delivery.

SECONDARY OUTCOMES:
Percentage of infants positive for HBsAg | At 9 months of life

OTHER OUTCOMES:
Percentage of women eligible for PAP who started TDF | At screening
Percentage of women eligible for PAP who completed TDF prophylaxis | up to 40 weeks of gestation
Percentage of women with adherence >90% at each study visit based on pill counts and self-report | from inclusion to delivery, max 40 weeks
Percentage of infants receiving HepB-BD | up to 9 months
Percentage of infants with a complete HepB vaccination schedule | up to 9 months
Percentage of women or infants with a serious adverse event (SAE) leading to death, or leading to treatment discontinuation up to delivery and Adverse Events of Special Interest | through study completion, an average of 27 months
Percentage of women who underwent liver disease assessment and factors associated with retention in care. | At 3 months postpartum
Percentage of women eligible for long-term TDF treatment | At 3 months post-partum
Accuracy (sensitivity, specificity, positive and negative predictive values) of the simplified score (HBcrAg-RDT & ALT) to predict eligibility for the long-term TDF treatment | At inclusion and 3 months after delivery
Communicative Health Literacy (COM_HL) on hepatitis B and related risks, empowerment, and health literacy among women and healthcare workers and factors associated | At 3-time points: inclusion, 6-8 weeks after delivery and 9 months after delivery
  Minimum total score = 5 Maximum total score = 25
  Low score:
  Indicates low communicative literacy.
  High score :
  Reflects a good ability to interact effectively in a healthcare context
Measures of the disclosure of HBV status among women and experience of sharing HBV status anf factors associated. | At 3-time points: inclusion, 6-8 weeks after delivery and 9 months after delivery
  Percentage of women who disclosed their HBV status to their partner and HBV disclosure score/moral support and discrimination scales
Percentage of partners and children who have been screened for HBV | At 3-time points: inclusion, 6-8 weeks after delivery and 9 months after delivery
Measures of perceived health and quality of life among women, the internalized stigma of mental illness and factors associated. | At 3-time points: inclusion, 6-8 weeks after delivery and 9 months after delivery
Acceptability for each strategy among healthcare workers, assessed using a scale adapted from Sekhon et al., 2022 to the intervention. | Before HCW training and at the end of the study (18-24 month after the study starts)
  Minimal total score= 0 Maximal total score= 100 Low score indicates low acceptability High score indicates high acceptability
. Measures of preferences of healthcare providers between the two strategies and associated factors | Before HCW training and at the end of the study (18-24 month after the study starts)
  Declared preferences of HCW between theoretical scenarios exhibiting various characteristics (time to get a diagnostic in minutes, cost for women in dollars, specificity and sensibility of the test in percentage)
.Cost per pregnant woman of the universal and of the targeted strategy, from the moment they are screened positive with the HBAgS (RDT) | until 9 months after delivery
  Costs will be estimated based on a societal approach, including all expenses for the healthcare system and the costs (direct and indirect) for the women and their households, and will be estimated using a dedicated data collection tool administrated during the duration of the project, relying on a micro-costing approach (see section 3.2.2 of the protocol, Health Economic Evaluation).
Incremental cost-effectiveness ratio (ICER) | At the end of follow_up after 27 months
  ICER wil be calculated as the difference in costs between the two strategies (incremental cost) divided by the difference in health benefits (infections avoided and mortality avoided between the two strategies). The ICER will be expressed as an additional cost (in dollars) per infection avoided.
  Lower ICER indicates greater cost-effectiveness of the assessed strategy.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier SEGERAL, Study Director — University Hospital, Geneva

IPD SHARING:
Plan to Share IPD: No